CLINICAL TRIAL: NCT01394861
Title: Endoscopic Submucosal Dissection (ESD)- Master Slave Robotic System - Human Study
Acronym: ESD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Collaborators: Nanyang Technological University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIG-GI2011-04
Record Dates: First submitted 2011-07-12; First posted 2011-07-15 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Endoscopic Submucosal Dissection
Keywords: Endoscopic Submucosal Dissection; ESD; EMR; Early Gastric Cancer; Flexible Endoscopic Robotic System; Master Slave Robot; Ease & Safety of ESD by Flexible Master Slave Robotic System
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ESD using MASTER Slave Robotic System (Experimental)
  Interventions: Device: ESD using Master Slave Robotic System

INTERVENTIONS:
Device: ESD using Master Slave Robotic System — Endoscopic submucosal dissection of early gastric cancer or broad sessile polyp using Master Slave Robotic System

SUMMARY:
The purpose of this study is to evaluate the feasibility, ease and safety of flexible endoscopic robotic system to treat early gastric cancer in humans.

DETAILED DESCRIPTION:
Aim:

To evaluate the feasibility and safety of Endoscopic Submucosal Dissection (ESD) using Master Slave Endoscopic Robotic System in humans.

Material and Methods:

To assess the feasibility and safety of ESD in humans, 3 patients with early gastric cancer or sessile polyp in the stomach with no evidence of involvement of deeper layer will be included in the study. The depth of involvement is evaluated by endoscopic ultrasound. An informed consent about the nature of the procedure, complications and the need for surgery will be explained to the patient. The master slave robot system (Human master robotic interface, telesurgical workstation and slave manipulator) and forward viewing therapeutic endoscope with 2 operating channels (GIF -2T160) will be used. The master controller controls the slave manipulator with electrical cables through a software interface. The slave manipulator in turn controls the end effectors (Monopolar 'L' hook and grasper) through cables passed through the two operating channels of the endoscope. The master slave robot system will be set up by the engineers from the Nanyang Technological University, Singapore. The endoscope will be connected to the high definition visual display and will be recorded throughout the procedure. Another high definition monitor will be set up for the surgeon/endoscopist who will control the MASTER at the console and the movements at the console will be continuously recorded. Monopolar electrocautery (ERBE) will be set up and tested. The settings for cutting and blend will be the same as used in the conventional ESD.

The therapeutic endoscope and the end effectors will be sterilised by immersing the scope in glutaraldehyde for 30 minutes before the procedure.

Patient will be kept fasting for 8 hours before the procedure. Under IV sedation, with the patient in left lateral position, end viewing diagnostic gastroscope is passed with an overtube. The lesion will be identified. Then the lesion will be marked by electrocautery (ERBE) all around. Then Gelofusine® (containing 4% succinylated gelatin, sodium hydroxide) stained with methylene blue will be injected submucosally under the lesion to create a cushion for ESD. Then IT knife is used for the mucosal cut all around the lesion. The double channel endoscope (GIF 2T160) will be exchanged through the overtube for the conventional endoscope after checking the system. Then submucosal dissection of the lesion will be performed, using the Master.

The data will be captured in the standard proforma for each patient. The endoscopic view and the external view of the MASTER will be recorded throughout the procedure.

Analysis - Efficacy and Safety outcomes:

The ease of the procedure (grasping, retraction, triangulation and complete excision), time required for mucosal cutting and submucosal dissection and completeness of the procedure will be analysed. Safety outcomes include intraoperative, immediate postoperative complications (bleeding, perforation) and the need for laparotomy will be assessed. Delayed Complications if any will be recorded for up to 30 days after the procedure.

Statistical Methodology:

As this is a pilot study, no sample size calculation was done. The aim is to perform the procedure in 3 subjects. Descriptive statistics will be used to describe safety data.

ELIGIBILITY:
Inclusion Criteria:

-Early Gastric Cancer or Gastric sessile polyp with dysplasia

Exclusion Criteria:

* Gastric Cancer with involvement of muscle layer
* Advanced Gastric cancer

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Ease of the procedure | 30 days
  The ease of the procedure (grasping, retraction, triangulation), time required for mucosal cutting and submucosal dissection

SECONDARY OUTCOMES:
Completeness of the Procedure | 30 days
  Completeness of the procedure is evaluated during the procedure by endoscopy and gross examination of the resected specimen followed by histopathological examination.
Immediate Procedure Related Complications | 30 days
  Bleeding or Perforation during and immediately after the procedure
Delayed Procedure Related Complications | 30 days
  Any complications (Delayed Bleeding or Perforation) related to the procedure up to thirty days post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Nageshwar Reddy Duvvuru, MD, DM, DSc, FAMS, FRCP, Principal Investigator — Asian Institute of Gastroenterology, India; Louis Soo Jay Phee, BEng, MEng, PhD, Principal Investigator — Nanyang Technological University
Locations (1):
- Asian Institute Of Gastroenterology India, Hyderabad, Andhra Pradesh, India